CLINICAL TRIAL: NCT04229849
Title: A Randomized, Open-label, Controlled, Multicenter Phase II Trial of Anrotenib Plus Toripalimab Versus Toripalimab for Following Treatment of Advanced Esophageal Squamous Cell Carcinoma After Chemotherapy Failure
Brief Title: Anrotenib Plus Toripalimab Versus Toripalimab in Patients With Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-GI-006
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anrotenib plus Toripalimab (Experimental): Anrotenib: 10 mg on day 1-14 orally repeated every 21 days; Toripalimab: 240 mg on day 1 intravenously repeated every 21 days; Until disease progression according to the RECIST 1.1 and irRECIST standard, intolerance of toxicity, withdrawal of informed consent from the subject, or tripleuriumab administration up to 2 years.
  Interventions: Drug: Anrotenib plus Toripalimab
- Toripalimab (Active Comparator): Toripalimab: 240 mg on day 1 intravenously repeated every 21 days; Until disease progression according to the RECIST 1.1 and irRECIST standard, intolerance of toxicity, withdrawal of informed consent from the subject, or tripleuriumab administration up to 2 years.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Anrotenib plus Toripalimab — Anrotenib: 10 mg on day 1-14 orally repeated every 21 days; Toripalimab: 240 mg on day 1 intravenously repeated every 21 days.
  Other Names: FOCUS V
  Arms: Anrotenib plus Toripalimab
Drug: Toripalimab — Toripalimab: 240 mg on day 1 intravenously repeated every 21 days.
  Arms: Toripalimab

SUMMARY:
The aim of this study is to investigate the efficacy and safety of anrotenib plus toripalimab in the treatment of advanced esophageal squamous cell carcinoma. In addition, the investigators will explore the possible mechanisms of anrotinib combined with toripalimab in advanced esophageal squamous cell carcinoma, and screen out biomarkers that can predict the efficacy of combination therapy.

DETAILED DESCRIPTION:
There is no standard recommendation for the treatment of advanced esophageal squamous cell cancer after chemotherapy failure. Anrotinib combined with triplizumab have showed synergistic effect in the tumor treatment, and they have demonstrated robust antitumor activity in the first-line treatment of advanced NSCLC with negative driving gene. However, there is no related report on the efficacy in the treatment of advanced esophageal squamous cell carcinoma. The aim of this study is to investigate the efficacy and safety of anrotenib plus toripalimab in the treatment of advanced esophageal squamous cell carcinoma. In addition, the investigators will explore the possible mechanisms of anrotinib combined with toripalimab in advanced esophageal squamous cell carcinoma, and screen out biomarkers that can predict the efficacy of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Confirmed esophageal squamous cell carcinoma patients by histopathological or cytopathological examinations.
* 2. Advanced esophageal squamous cell carcinoma patients with progression after chemotherapy of taxol and/or platinum or fluorouracil.
* 3. According to the evaluation criteria of solid tumor efficacy (RESIST 1.1), there should be at least one measurable lesion (empty organs such as esophagus and stomach cannot be taken as the measurable lesion), and the measurable lesion should not have received local treatment such as radiotherapy (the lesion located in the previous radiotherapy area is also selected as the target lesion if the lesion progression is confirmed).
* 4. A histological specimen can be provided for secondary testing.
* 5. ≥18 years old, male or female.
* 6. ECOG performance status 0-1.
* 7. Life expectancy ≥ 12 weeks.
* 8. The main organ function meets the following criteria within 7 days before treatment:

  1. Blood routine examination criteria (without blood transfusion within 14 days): hemoglobin (HB) ≥ 90g/L, the absolute value of neutrophils (ANC) ≥ 1.5 x 10^9/L, platelet (PLT) ≥ 80 x 10^9/L.
  2. Biochemical examinations must meet the following criteria: total bilirubin (TBIL) ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x ULN, serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance (CCR) ≥ 60 mL/min.
  3. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).
* 9. Fertile men and women must use effective contraception during the study period and within 6 months after the end of the study.
* 10. The patient volunteered to participate in the study and signed an informed consent form.

Exclusion Criteria:

* 1.Patients exceeding or currently suffering from other malignant tumors within 5 years, except for cervical cancer in site, non-melanoma skin cancer and superficial bladder tumors (Ta (non-invasive tumor), Tis (in situ carcinoma), and T1 (tumor infiltrating basement membrane)); Patients with rapid progress within 3 months.
* 2. History of gastrointestinal perforation and/or fistula within 6 months prior to the first administration.
* 3. Esophageal lesion obviously invading the adjacent organs (major arteries or trachea), resulting in a higher risk of bleeding or fistula.
* 4. Received any of the following treatment:

  1. Previous treatment with anti-PD-1 antibodies or anti-PD-L1 antibodies;
  2. Received any experimental drug within 4 weeks prior to the first administration of the study drug;
  3. Enroll in another clinical study, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up;
  4. Receive the last dose of anticancer therapy (including radiotherapy, etc.) within 4 weeks before the first administration of the study drug;
  5. Patients who need to be given corticosteroids (the equivalent dose of > 10 mg prednisone per day) or other immunosuppressants for systemic treatment within 2 weeks prior to the first use of the study drug, except the use of corticosteroids for esophageal local inflammation and the prevention of allergies, nausea and vomiting. In the absence of active autoimmune disease, inhaled or topical corticosteroid of an equivalent dose of > 10mg prednisone per day is permitted;
  6. Received an anti-tumor vaccine or received a live vaccine within 4 weeks prior to the first administration of the study drug
  7. Received major surgery or severe trauma within 4 weeks prior to first administration of the study drug.
* 5. History of immunodeficiency disease, including HIV positive and other acquired or congenital immunodeficiency diseases, or history of organ transplantation allogeneic bone marrow transplantation.
* 6. Toxicity of previous antitumor treatment did not return to the level ≤NCI CTC AE V5.0 grade 1 (except alopecia) or to the level specified in the inclusion/exclusion criteria.
* 7. History of allergy to monoclonal antibody or the ingredients of the study drug.
* 8. Significantly malnourished patients. Exclusion is performed if the patient is receiving intravenous fluids or is required to be hospitalized for continuous infusion therapy. Patients with good nutrition control ≥ 28 days can be enrolled before randomization.
* 9. Any severe and/or uncontrolled disease, including:

  1. Patients with hypertension whose blood pressure can't be well controlled by antihypertensive drugs (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg);
  2. Grade 1 or higher myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥ 480 ms) or grade 2 and above congestive heart failure according to New York Heart Association (MYHA) classification;
  3. Severe or uncontrolled disease or active infection (≥ NCI CTC AE V5.0 grade 2), which the investigators believe may increase the risk associated with patient participation and drug administration;
  4. Renal failure requiring hemodialysis or peritoneal dialysis;
  5. Patients of diabetes who have poor glycemic control (fasting blood glucose (FBG) > 10 mmol/L);
  6. Urine routine showed urinary protein ≥ 2 + and 24-hour urine protein quantitation > 1.0 g;
  7. Patients of seizures requiring treatment.
* 10. Any bleeding event ≥ NCI CTC AE V5.0 grade 3 or unhealed wounds, ulcers or fractures in 4 weeks prior to enrollment.
* 11. Arterial/venous thrombosis events within 3 months, such as cerebrovascular accidents (including transient ischemic attacks), deep venous thrombosis and pulmonary embolism.
* 12. Active autoimmune diseases or the history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Except patients with vitiligo or childhood asthma/allergies that have been cured and do not require any intervention as adults, autoimmune hypothyroidism treated with a stable dose of thyroid replacement hormone, type 1 diabetes using a steady dose of insulin.
* 13. History of interstitial pulmonary disease (excluding radiation pneumonia without hormone therapy) and non-infectious pneumonia.
* 14. Patients with active pulmonary tuberculosis infection found by medical history or CT examination, or with a history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or with a history of active pulmonary tuberculosis infection more than 1 year prior to enrollment but without formal treatment.
* 15. Patients with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL) and hepatitis C (HCV-RNA higher than the lower limit of the assay).
* 16. Patients may have other factors that cause them to be forced to terminate the study, such as other serious diseases (including mental illness) that require combined treatment, serious abnormalities in laboratory test, and family or social factors, which may affect the safety of patients or the collection of experimental data.
* 17. Patients with brain metastases.
* 18. Woman who is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  From the first day of treatment to death or last survival confirm date

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 years
  From the first day of treatment until the date of first documented progression or date of death from any cause
Objective Response Rate (ORR) | up to 2 years
  To compare objective response rate of the two arms from date of anti-cancer therapy until progression
Disease Control Rate (DCR) | up to 2 years
  To compare disease control rate of the two arms from date of anti-cancer therapy until progression
Number of Participants with Treatment-related Adverse Events Treatment-related adverse events | up to 2 years
  Number of Participants with Treatment-related Adverse Events Treatment-related adverse events will be assessed by NCI CT CAE v5.0
Assessment of Health-related quality of life | up to 2 years
  Quality of Life Questionnaire (QLQ-C30) will be evaluated since treatment begins. At the end of the trail, the differences between the two indicators will be compared with Mixed-effects model repeated measures (MMRM), where the baseline is scored as a covariant and the treatment group as a fixed variable. In addition, the baseline values of the two scores, the value of each visit, and the change value of the baseline will be statistically described.

CONTACTS AND LOCATIONS:
Overall Officials: Baoxia He, Study Director — Henan Cancer Hospital/The affiliated Cancer Hospital of Zhengzhou University